CLINICAL TRIAL: NCT07157241
Title: Effect of Omega-3 Supplements on Stress, Anxiety, Depression, Memory and Sleep Quality Among Saudi Adults: A Double-Blind Placebo Randomized Controlled Trial
Brief Title: Effect of Omega-3 Supplements on Stress, Anxiety, Depression, Memory and Sleep Quality Among Saudis
Acronym: OSADMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Wedad Azhar, Dr. Wedad Azhar, Assistant Professor, Umm Al-Qura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HAPO-02-K-012-2021-11-832; UmmAlQuraU (Other: Umm Al-Qura University)
Record Dates: First submitted 2025-07-11; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Healthy Adults; Anxiety; Depression; Sleep Quality; Everyday Memory; Psychological Distress
Keywords: omega-3; stress; anxiety; mental distress; Psychological Distress; healthy adults; depression; sleep Quality; Everyday Memory; Saudi Arabia
MeSH Terms: conditions — Anxiety Disorders; Depression; Sleep Initiation and Maintenance Disorders | interventions — Methods; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Placebo Comparator): corn oil 400 mg capsule a day for for three months
  Interventions: Dietary Supplement: Control group (placebo)
- intervention group (Experimental): mega-3 capsules with a concentration of 1000 mg/day for three months (NOW Foods- Ultra omega-3 500 EPA/250 DHA).
  Interventions: Dietary Supplement: Intervention

INTERVENTIONS:
Dietary Supplement: Intervention — omega-3 capsules with a concentration of 1000 mg/day for three months (NOW Foods- Ultra omega-3 500 EPA/250 DHA).
  Arms: intervention group
Dietary Supplement: Control group (placebo) — corn oil capsule /day for 3 months
  Arms: Control

SUMMARY:
This study looked at whether taking omega-3 supplements can help reduce stress, anxiety, depression, and improve memory and sleep quality in Saudi adults who feel highly stressed or anxious. Omega-3 is a healthy fat found in fish oil that may help the brain and mood.

A total of 64 adults took part. They were randomly split into two groups. One group took omega-3 capsules (500 mg EPA + 250 mg DHA) every day for three months. The other group took a placebo (an inactive oil). Neither the participants nor the researchers knew who was taking which capsules to keep the study fair.

Before and after the three months, all participants completed simple questionnaires about their stress, anxiety, depression, sleep, and everyday memory.

The results showed that people who took omega-3 had lower stress, anxiety, and depression scores and reported better sleep quality and memory compared to those who took the placebo.

This suggests that taking omega-3 supplements may help improve mental wellbeing and sleep in people with high stress and anxiety.

DETAILED DESCRIPTION:
Psychological stress, anxiety, depression, memory difficulties, and poor sleep quality are common issues that affect many adults and can lower overall health and quality of life. Although pharmaceutical treatments exist, they often come with side effects and may not work for everyone. Nutritional approaches, such as omega-3 polyunsaturated fatty acid (PUFA) supplementation, have gained interest due to their possible neuroprotective, anti-inflammatory, and mood-regulating effects.

This study investigated the impact of daily omega-3 supplementation (500 mg EPA + 250 mg DHA) for three months compared with placebo in Saudi adults with high levels of stress and anxiety. Validated tools - including the Perceived Stress Scale (PSS), Generalized Anxiety Disorder-7 (GAD-7), Patient Health Questionnaire-9 (PHQ-9), Everyday Memory Questionnaire (EMQ), and sleep quality scales (PSQI, ESS) - were used to assess changes before and after the intervention.

The trial used a randomized, double-blind, placebo-controlled design. Adherence was monitored through daily communication and monthly capsule counts. Results indicated significant improvements in stress, anxiety, depression, memory, and sleep quality for participants who received omega-3 compared with those who received placebo. Statistical analyses showed strong effect sizes and predictive relationships between baseline measures and outcomes.

This research highlights the potential role of omega-3 supplementation as a supportive strategy for mental wellbeing and sleep improvement. Further studies are needed to explore individual responses and underlying biological mechanisms.

ELIGIBILITY:
Inclusion Criteria:

high psychological distress did not take any omega-3 supplements for the last 6 month

-

Exclusion Criteria:

* younger than 18 pregnant breastfeeding anyone with supplements and chronic diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-02-27 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
Change from the baseline for the following scales: Perceived Stress General Anxiety Disorder-7 Depression Level measured using PHQ-9 Sleep Quality Daytime sleepiness and sleep disorders Memory failure in everyday life. | Baseline and 3 months after intervention
  Primary Outcome Measures:
  1. Change in Perceived Stress Perceived Stress Scale (0-40, higher = more stress). Self-reported at baseline and 3 months.
  2. Change in Anxiety Level Generalized Anxiety Disorder-7 (0-21, higher = more anxiety). Self-reported at baseline and 3 months.
  3. Change in Depression Level Patient Health Questionnaire-9 (0-27, higher = more depression). Self-reported at baseline and 3 months.
  4. Change in Sleep Quality Pittsburgh Sleep Quality Index (0-21, higher = poorer sleep quality). Self-reported at baseline and 3 months.
  5. Change in Daytime Sleepiness Epworth Sleepiness Scale (0-24, higher = more sleepiness). Self-reported at baseline and 3 months.
  6. Change in Everyday Memory Failures Everyday Memory Questionnaire (0-25, higher = more frequent memory failures). Self-reported at baseline and 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Qadhi, Ph.D, Study Director — Umm Al-Qura University
Locations (1):
- university of Umm Al-Qura, Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
There are no plans to share IPD to protect participant confidentiality. Study results are published in summary form only.

REFERENCES:
- [Derived] Azhar W, Qadhi A, Abusudah W, Ghabashi M, Aljaadi AM, Alyamani R, Awlya O, Almohmadi N, Alsemeri A, Felemban A, Alturki G, Almatrafi L, Zafarani R, Kamfar Y, Azzeh F, Ghafouri K. The effects of Omega-3 supplementation on stress, anxiety, depression, sleep quality, and everyday memory in individuals with psychological distress: A randomized, double-blind, placebo-controlled trial. J Affect Disord. 2026 Apr 15;399:121055. doi: 10.1016/j.jad.2025.121055. Epub 2025 Dec 27. PMID 41461240